CLINICAL TRIAL: NCT04913610
Title: A Phase-II, Randomised, Double-blind, Parallel-group, Proof-of-concept Trial to Investigate ABBV-4083 Given for 7 or 14 Days or in Combination With Albendazole in Subjects With Onchocerca Volvulus Infection, Comprising: Part 1 to Investigate Safety, Tolerability, Efficacy for Dose-Ranging and Pharmacokinetics; Part 2 to Investigate Efficacy of Selected Doses, Safety, Tolerability and Pharmacokinetics
Brief Title: Study to Assess Adverse Events, Change in Disease Activity and How Oral ABBV-4083 Capsules When Given Alone or In Combination With Albendazole Capsules Moves in The Body of Adult Participants With Onchocerca Volvulus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Collaborators: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B18-894; DNDi-TYL-01 (Other: DNDi)
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Onchocerciasis
Keywords: Onchocerciasis; Onchocerca volvulus; River blindness; ABBV-4083; Tylamac
MeSH Terms: conditions — Onchocerciasis; Onchocerciasis, Ocular | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 pbo for 7 days (Experimental): Participants received ABBV-4083 400 mg administered orally as capsules plus placebo capsules for albendazole for 7 days followed by placebo capsules for ABBV-4083 for 7 days.
  Interventions: Drug: ABBV-4083; Drug: Placebo for ABBV-4083; Drug: Placebo for Albendazole
- Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 400 mg for 7 days (Experimental): Participants received ABBV-4083 400 mg administered orally as capsules plus placebo capsules for albendazole for 7 days followed by ABBV-4083 400 mg administered orally as capsules for 7 days.
  Interventions: Drug: ABBV-4083; Drug: Placebo for Albendazole
- Part 1: ABBV-4083 400 mg + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days (Experimental): Participants received ABBV-4083 400 mg administered orally as capsules plus albendazole 400 mg capsules for 7 days followed by placebo capsules for ABBV-4083 for 7 days.
  Interventions: Drug: ABBV-4083; Drug: Placebo for ABBV-4083; Drug: Albendazole
- Part 1: ABBV-4083/albendazole 400 mg 3 d; ABBV-4083 400 mg/albendazole pbo 4 d; ABBV-4083 pbo 7 d (Experimental): Participants received ABBV-4083 400 mg administered orally as capsules plus albendazole 400 mg capsules for 3 days followed by ABBV-4083 400 mg and placebo capsules for albendazole for 4 days followed by placebo capsules for ABBV-4083 for 7 days.
  Interventions: Drug: ABBV-4083; Drug: Placebo for ABBV-4083; Drug: Albendazole; Drug: Placebo for Albendazole
- Part 1: ABBV-4083 pbo + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days (Experimental): Participants received placebo for ABBV-4083 administered orally as capsules plus albendazole 400 mg capsules for 7 days followed by placebo capsules for ABBV-4083 for 7 days.
  Interventions: Drug: Placebo for ABBV-4083; Drug: Albendazole

INTERVENTIONS:
Drug: ABBV-4083 — Oral Capsule
  Other Names: Tylamac
  Arms: Part 1: ABBV-4083 400 mg + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 400 mg for 7 days; Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083/albendazole 400 mg 3 d; ABBV-4083 400 mg/albendazole pbo 4 d; ABBV-4083 pbo 7 d
Drug: Placebo for ABBV-4083 — Oral Capsule
  Arms: Part 1: ABBV-4083 400 mg + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083 pbo + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083/albendazole 400 mg 3 d; ABBV-4083 400 mg/albendazole pbo 4 d; ABBV-4083 pbo 7 d
Drug: Albendazole — Oral encapsulated tablets
  Other Names: Zentel
  Arms: Part 1: ABBV-4083 400 mg + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083 pbo + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083/albendazole 400 mg 3 d; ABBV-4083 400 mg/albendazole pbo 4 d; ABBV-4083 pbo 7 d
Drug: Placebo for Albendazole — Oral Capsule
  Arms: Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 400 mg for 7 days; Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 pbo for 7 days; Part 1: ABBV-4083/albendazole 400 mg 3 d; ABBV-4083 400 mg/albendazole pbo 4 d; ABBV-4083 pbo 7 d

SUMMARY:
Onchocerciasis is a major public health problem in affected countries that causes disease-induced disability, and overall loss of economic productivity. The purpose of this study is to determine how safe and effective ABBV-4083 in combination with albendazole is in treating participants with Onchocerciasis.

ABBV-4083 is an investigational drug being developed for the treatment of onchocerciasis. This study is conducted in 2 parts. In part 1, participants are randomly assigned to 1 of 5 groups, called treatment arms to determine the most efficient treatment combination. Each group receives a different treatment. In part 2, participants are randomly assigned to 1 of 4 treatment arms. Approximately 444 or 486 adult participants with a diagnosis of onchocerciasis will be enrolled in approximately 2 sites in Democratic Republic of Congo.

Participants in Part 1 will receive different treatment combinations of ABBV-4083 and/or albendazole and/or matching placebo capsules for 14 days. Participants in Part 2 will receive the most effective treatment combination(s) determined in Part 1 for 14 days followed by ivermectin or matching placebo capsules at Month 6; duration of treatment is 24 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests and checking for side effects.

DETAILED DESCRIPTION:
The study was terminated at the conclusion of Part 1, and Part 2 of the study was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Onchocerca volvulus infection at time of Screening:

  * Presence of at least one excisable subcutaneous nodule/ onchocercoma detected on palpation;
  * O. volvulus infection diagnosed by skin snip method: documented mfpositivity on skin assessment on at least 2 out of 4 skin snips.
* Body weight > 40 kg at Screening.
* For women of child-bearing potential, acceptance of the requirement to use a highly effective form of birth control from Day 0 until at least 1 month after the final intake of study drug (Part 1: day 43; Part 2: 1 month after the administration of ivermectin or matching placebo at the Month 6 visit). Choice of birth control method must be clearly documented.

Exclusion Criteria:

* Participation in any studies other than purely observational studies within 3 months prior to Screening, or during the trial, or within 5 times the half-life of the drug tested in the previous clinical trial or is currently in the follow-up period for any clinical trial.
* Any vaccination within 4 weeks prior to investigational medicinal product (IMP) administration.
* Acute infection and/or febrile illness requiring therapy within 14 days prior to IMP administration.
* Administration of medication or herbal preparations as follows:

  * Administration of any medication (with the exception of diclofenac, paracetamol, ibuprofen and aspirin) or herbal preparation within 14 days prior to IMP administration;
  * Use of strong CYP3A inhibitors or inducers including but not limited to ritonavir, ketoconazole, rifampicin, phenytoin, phenobarbital, carbamazepine, cimetidine within 14 days or 10 half-lives, whichever is longer, prior to IMP administration;
  * Use of other drugs known to interact with albendazole i.e. praziquantel, theophylline or dexamethasone, within 14 days or 10 half-lives, whichever is longer, prior to IMP administration;
  * Antifilarial therapies, or medication that may have an antifilarial effect.
* Requirement for and inability to avoid ivermectin during the first 6 months after IMP administration. Requirement for albendazole during the first 28 days after IMP administration or more than one dose per year thereafter given in MDA.
* Presence of any of the following at Screening, that could interfere with the objectives of the trial or the safety of the participant, in the opinion of the Investigator:

  * Clinically significant abnormal physical and/or neurological examination or laboratory findings;
  * Any clinically significant medical condition. Including, but not limited to significant acute or chronic liver or kidney condition or cardiovascular disease, active infection, current or previous epilepsy, known human immunodeficiency virus infection, disclosed by review of medical history or concomitant medication.
* Ophthalmological history or conditions that could interfere with the objectives of the trial or compromise the safety of the subject in the opinion of the Investigator, assessed at Screening.
* History of drug or alcohol abuse within 6 months prior to IMP administration.
* Use of alcohol within 48 hours and/or use of drugs of abuse within 15 days before IMP administration.
* Clinically significant history of cardiac abnormality, and/or relevant pathological abnormalities in the ECG in the screening period.
* Abnormal laboratory test results at Screening.
* History of severe drug allergy, non-allergic drug reactions, severe adverse reaction to any drug, or multiple drug allergies.
* Known hypersensitivity to any ingredient of the IMPs, including the active ingredient of ABBV-4083, macrolides, albendazole or to ivermectin or to any medication used during the study.
* Blood donation within 8 weeks prior to Screening or blood transfusion received within 1 year prior to Screening.
* Coincidental infection with high Loa loa load at Screening.
* Current hyperreactive onchodermatitis or severe manifestation due to onchocerciasis.
* Any other past or current condition that the Investigator feels would exclude the participant from the study or place the subject at undue risk.
* For women of child-bearing potential: pregnant, based on date of last menstrual period, and pregnancy test prior to first intake of IMP, or breastfeeding.
* Unwilling or unable to comply with the requirements of the study protocol for the entire duration of the study, in the opinion of the Investigator.
* Unable to participate in the study as per local law, if applicable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- Democratic Republic of the Congo (2):
  - Hôpital Général de Référence de Kimpese, Kimpese, Bas-Congo Province
  - Hôpital Général de Référence de Masi-Manimba, Masi-Manimba, Kwilu

IPD SHARING:
Plan to Share IPD: No
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 153 participants were randomized, of which 151 received study drug (Intention-to-Treat, ITT; Safety population).
Period: Randomized Participants
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Started | 31 | 31 | 30 | 30 | 31
Completed | 31 | 31 | 29 | 29 | 31
Not Completed | 0 | 0 | 1 | 1 | 0
Not completed — Did Not Receive Treatment | 0 | 0 | 1 | 1 | 0
Period: Treated (ITT & Safety Population)
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Started | 31 | 31 | 29 | 29 | 31
Completed | 30 | 31 | 29 | 29 | 30
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population includes all randomized participants who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Total
Number analyzed (Participants) | 31 | 31 | 29 | 29 | 31 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (10.36) | 37.1 (11.73) | 40.1 (12.08) | 38.7 (10.78) | 38.5 (12.34) | 39.6 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 0 | 4 | 6 | 16
  Male | 29 | 27 | 29 | 25 | 25 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was not collected from any participant.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 31 | 31 | 29 | 29 | 31 | 151
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body weight [Mean (Standard Deviation); unit: kilograms] | 53.55 (7.03) | 50.98 (6.04) | 53.48 (7.12) | 52.38 (6.42) | 49.77 (6.96) | 52.01 (6.80)
Number of operable sites with onchocercomata [Mean (Standard Deviation); unit: sites] | 1.5 (0.72) | 1.6 (0.67) | 1.6 (0.74) | 1.6 (1.02) | 1.5 (0.68) | 1.5 (0.76)
Number of palpated onchocerca nodules [Mean (Standard Deviation); unit: nodules] | 1.7 (0.83) | 1.7 (0.70) | 1.7 (1.03) | 1.8 (1.15) | 1.7 (0.93) | 1.7 (0.92)
Skin microfilarial density [Mean (Standard Deviation); unit: mf/mg of skin] | 8.22 (12.25) | 26.55 (33.06) | 20.60 (35.52) | 19.45 (34.97) | 16.59 (25.81) | 18.23 (29.71)
Number of previous ivermectin rounds [Mean (Standard Deviation); unit: rounds] | 0.4 (0.71) | 0.0 (0.18) | 0.4 (0.87) | 0.3 (0.59) | 0.2 (0.67) | 0.3 (0.65)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Live Female Adult Worms Without Wolbachia at Month 6 as Assessed By Immunohistology of Nodules
Description: The Wolbachia endobacteria status of each live female adult worm was determined by immunohistology of nodules collected after nodulectomy at the Month 6 visit.
Time Frame: At Month 6
Population: Per protocol population: all ITT participants who had nodulectomy at Month 6 (ND6M) with live female adult worms, who completed treatment, and who did not take prohibited medication(s) during the study
Measure: Number (95% Confidence Interval); unit: Percentage of worms without Wolbachia
Units Other Than Participants: Live female adult worms with data
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 22 | 23 | 22 | 21 | 20
Number analyzed (Live female adult worms with data) | 84 | 87 | 82 | 90 | 77
Percentage of worms without Wolbachia | 6.0 [2.6 to 13.2] | 2.3 [0.6 to 8.0] | 0.0 [0.0 to 4.5] | 0.0 [0.0 to 4.1] | 2.6 [0.7 to 9.0]

2. Secondary Outcome: Part 1: Percentage of Live Female Adult Worms With Only Degenerated Embryos in the Uterus Per Participant at Month 6
Description: The percentage of live female adult worms with only degenerated embryos in the uterus per participant was determined after nodulectomy at the Month 6 visit.
Time Frame: At Month 6
Population: Intention-to-treat (ITT) population who had live female adult worms that contained either normal embryos, degenerated embryos, or both
Measure: Mean (Standard Deviation); unit: Percentage of worms per participant
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 19 | 20 | 19 | 18 | 16
Percentage of worms per participant | 0.48 (2.086) | 7.67 (18.420) | 9.82 (19.578) | 7.59 (23.813) | 10.16 (18.064)
Statistical Analysis 1: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 pbo for 7 days (Arm A) versus Part 1: ABBV-4083 pbo + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days (Arm E); Test type: Other; p = 0.036, Mann-Whitney U test; The p-value is for the pairwise comparison of Arm A to Arm E using the Mann-Whitney U test for the percentage per participant
Statistical Analysis 2: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; Part 1: ABBV-4083 400 mg + albendazole pbo for 7 days, then ABBV-4083 400 mg for 7 days (Arm B) versus Part 1: ABBV-4083 pbo + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days (Arm E); Test type: Other; p = 0.530, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm B to Arm E using the Mann-Whitney U test for the percentage per participant
Statistical Analysis 3: Comparison: Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; Part 1: ABBV-4083 400 mg + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days (Arm C) versus Part 1: ABBV-4083 pbo + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days (Arm E); Test type: Other; p = 0.852, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm C to Arm E using the Mann-Whitney U test for the percentage per participant
Statistical Analysis 4: Comparison: Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; Part 1: ABBV-4083/albendazole 400 mg 3 d; ABBV-4083 400 mg/albendazole pbo 4 d; ABBV-4083 pbo 7 d (Arm D) versus Part 1: ABBV-4083 pbo + albendazole 400 mg for 7 days, then ABBV-4083 pbo for 7 days (Arm E); Test type: Other; p = 0.366, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm D to Arm E using the Mann-Whitney U test for the percentage per participant

3. Secondary Outcome: Part 1: Percentage of Live Female Adult Worms Out of All Female Adult Worms Per Participant at Month 6
Description: The percentage of live female adult worms out of all female adult worms per participant was determined after nodulectomy at the Month 6 visit.
Time Frame: At Month 6
Population: Intention-to-treat (ITT) population who had female adult worms
Measure: Mean (Standard Deviation); unit: Percentage of worms per participant
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 22 | 26 | 24 | 22 | 22
Percentage of worms per participant | 84.27 (19.904) | 77.74 (32.445) | 78.03 (29.811) | 79.37 (27.013) | 79.52 (30.496)
Statistical Analysis 1: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.869, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm A to Arm E using the Mann-Whitney U test for the percentage per participant
Statistical Analysis 2: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.973, Mann-Whitney U test — [p-value comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.744, Mann-Whitney U test — [p-value comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.794, Mann-Whitney U test — [p-value comment as in outcome 2, analysis 4]

4. Secondary Outcome: Part 1: Percentage of Participants Without Microfilariae in Nodular Tissue at Month 6
Description: The absence of microfilariae in nodular tissue per participant was determined after nodulectomy at the Month 6 visit.
Time Frame: At Month 6
Population: Intention-to-treat (ITT) population who had post-baseline values at Month 6
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 22 | 26 | 24 | 22 | 23
Percentage of participants | 22.7 | 26.9 | 41.7 | 31.8 | 30.4
Statistical Analysis 1: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.559, Chi-square test — The p-value is for the pairwise comparison of Arm A to Arm E using the using the Chi-square test for the binary response per participant
Statistical Analysis 2: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.786, Chi-square test — The p-value is for the pairwise comparison of Arm B to Arm E using the using the Chi-square test for the binary response per participant
Statistical Analysis 3: Comparison: Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.423, Chi-square test — The p-value is for the pairwise comparison of Arm C to Arm E using the using the Chi-square test for the binary response per participant
Statistical Analysis 4: Comparison: Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.920, Chi-square test — The p-value is for the pairwise comparison of Arm D to Arm E using the using the Chi-square test for the binary response per participant

5. Secondary Outcome: Part 1: Percentage of Participants Without Skin Microfilariae at Month 3
Description: The presence or absence of microfilariae in skin was determined at the Month 3 visit.
Time Frame: At Month 3
Population: Intention-to-treat (ITT) population who had post-baseline values at Month 3
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 31 | 31 | 28 | 28 | 30
Percentage of participants | 3.2 | 3.2 | 3.6 | 3.6 | 3.3
Statistical Analysis 1: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.981, Chi-square test — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.981, Chi-square test — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.960, Chi-square test — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.960, Chi-square test — [p-value comment as in outcome 4, analysis 4]

6. Secondary Outcome: Part 1: Percentage of Participants Without Skin Microfilariae at Month 6
Description: The presence or absence of microfilariae in skin was determined at the Month 6 visit.
Time Frame: At Month 6
Population: Intention-to-treat (ITT) population who had post-baseline values at Month 6
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 27 | 28 | 28 | 25 | 28
Percentage of participants | 0 | 0 | 0 | 0 | 7.1
Statistical Analysis 1: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.157, Chi-square test — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.150, Chi-square test — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.150, Chi-square test — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.173, Chi-square test — [p-value comment as in outcome 4, analysis 4]

7. Secondary Outcome: Part 1: Mean Within-Participant Change From Baseline in Skin Microfilarial Density at Month 3
Description: Skin microfilarial density is defined as the mean number of microfilariae/mg of skin per participant.
Time Frame: Baseline, Month 3
Population: Intention-to-treat (ITT) population who had values at Baseline and Month 3
Measure: Mean (Standard Deviation); unit: Mean number of microfilariae/mg of skin
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 31 | 31 | 28 | 28 | 30
Mean number of microfilariae/mg of skin | -0.44 (5.576) | -7.99 (16.180) | 2.43 (13.148) | 1.36 (12.189) | -1.03 (10.787)
Statistical Analysis 1: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.619, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm A to Arm E using the Mann-Whitney U test for the change from baseline in skin microfilarial density per participant
Statistical Analysis 2: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.194, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm B to Arm E using the Mann-Whitney U test for the change from baseline in skin microfilarial density per participant
Statistical Analysis 3: Comparison: Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.518, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm C to Arm E using the Mann-Whitney U test for the change from baseline in skin microfilarial density per participant
Statistical Analysis 4: Comparison: Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.652, Mann-Whitney U test — The p-value is for the pairwise comparison of Arm D to Arm E using the Mann-Whitney U test for the change from baseline in skin microfilarial density per participant

8. Secondary Outcome: Part 1: Mean Within-Participant Change From Baseline in Skin Microfilarial Density at Month 6
Description: Skin microfilarial density is defined as the mean number of microfilariae/mg of skin per participant.
Time Frame: Baseline, Month 6
Population: Intention-to-treat (ITT) population who had values at Baseline and Month 6
Measure: Mean (Standard Deviation); unit: Mean number of microfilariae/mg of skin
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 27 | 28 | 28 | 25 | 28
Mean number of microfilariae/mg of skin | -0.19 (6.330) | 5.55 (24.293) | -1.19 (32.856) | -2.72 (19.769) | -1.67 (14.223)
Statistical Analysis 1: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.386, Mann-Whitney U test — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.279, Mann-Whitney U test — [p-value comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.385, Mann-Whitney U test — [p-value comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d vs Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.755, Mann-Whitney U test — [p-value comment as in outcome 7, analysis 4]

9. Secondary Outcome: Part 1: Percentage of Nodules That Contain at Least 1 Live Female Adult Worm Without Wolbachia Assessed by PCR at Month 6
Description: The Wolbachia endobacteria status of each live female adult worm was determined by PCR of nodules collected after nodulectomy at the Month 6 visit.
Time Frame: At Month 6
Population: Intention-to-treat (ITT) population who had live female adult worms
Measure: Number; unit: Percentage of nodules
Units Other Than Participants: Nodules w/live female adult worms + data
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days
Number analyzed (Participants) | 22 | 26 | 24 | 22 | 22
Number analyzed (Nodules w/live female adult worms + data) | 26 | 32 | 21 | 32 | 17
Percentage of nodules | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were collected from the time informed consent was signed through the end of the study. Median time on follow-up was 201 days for Arms A, B, C, and all participants randomized to receive ABBV-4083; 210 days for Arm D; and 213 days for Arm E.
Groups:
- Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days (A): Participants randomized to receive ABBV-4083 400 mg administered orally as capsules plus placebo capsules for albendazole for 7 days followed by placebo capsules for ABBV-4083 for 7 days.
- Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days (B): Participants randomized to receive ABBV-4083 400 mg administered orally as capsules plus placebo capsules for albendazole for 7 days followed by ABBV-4083 400 mg administered orally as capsules for 7 days.
- Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (C): Participants randomized to receive ABBV-4083 400 mg administered orally as capsules plus albendazole 400 mg capsules for 7 days followed by placebo capsules for ABBV-4083 for 7 days.
- Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d(D): Participants randomized to receive ABBV-4083 400 mg administered orally as capsules plus albendazole 400 mg capsules for 3 days followed by ABBV-4083 400 mg and placebo capsules for albendazole for 4 days followed by placebo capsules for ABBV-4083 for 7 days.
- Participants Randomized to Receive ABBV-4083 (Arms A, B, C, and D): All participants who were randomized to receive ABBV-4083
- Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (E): Participants randomized to receive placebo for ABBV-4083 administered orally as capsules plus albendazole 400 mg capsules for 7 days followed by placebo capsules for ABBV-4083 for 7 days.
Arm/Group | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days (A) | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days (B) | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (C) | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d(D) | Participants Randomized to Receive ABBV-4083 (Arms A, B, C, and D) | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (E)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/30 | 0/122 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/31 | 2/30 | 0/30 | 4/122 | 4/31
Other Adverse Events (participants affected / at risk) | 14/31 | 9/31 | 13/30 | 10/30 | 46/122 | 14/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days (A) (N=31) | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days (B) (N=31) | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (C) (N=30) | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d(D) (N=30) | Participants Randomized to Receive ABBV-4083 (Arms A, B, C, and D) (N=122) | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (E) (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RETINAL VEIN OCCLUSION (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIODONTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 Pbo for 7 Days (A) (N=31) | Part 1: ABBV-4083 400 mg + Albendazole Pbo for 7 Days, Then ABBV-4083 400 mg for 7 Days (B) (N=31) | Part 1: ABBV-4083 400 mg + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (C) (N=30) | Part 1: ABBV-4083/Albendazole 400 mg 3 d; ABBV-4083 400 mg/Albendazole Pbo 4 d; ABBV-4083 Pbo 7 d(D) (N=30) | Participants Randomized to Receive ABBV-4083 (Arms A, B, C, and D) (N=122) | Part 1: ABBV-4083 Pbo + Albendazole 400 mg for 7 Days, Then ABBV-4083 Pbo for 7 Days (E) (N=31)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 7 (7) | 2 (2) | 16 (16) | 2 (2)
EYE PRURITUS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
VISUAL FIELD DEFECT (Eye disorders) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 6 (7) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
MALARIA (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 9 (9) | 6 (6)
SCHISTOSOMIASIS BLADDER (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 7 (7) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A multisite publication of the results is made prior to any publication based on results obtained by a specific site. Written publications or oral presentations that include all or part of the results must be sent to DNDi for review and comment at least 28 days prior to the planned date of publication/presentation. In addition, publication/presentation of results will be delayed for a further 90 days in the event that DNDi wishes to protect the results by patent application or other means.

DOCUMENTS (2):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT04913610/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT04913610/SAP_001.pdf